CLINICAL TRIAL: NCT06119789
Title: The MATRIX Clinical Studies of Precision Cancer Therapy for Rare Cancers
Brief Title: Precision Cancer Therapy in Rare Cancers
Acronym: MATRIX-Rare
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); University Hospital of North Norway (Other); StOlavs Hospital (Unknown); Nordlandssykehuset HF (Other); Helse Nord-Trøndelag HF (Other); Sorlandet Hospital HF (Other Government); Møre og Romsdal Hospital Trust (Other); The Hospital of Vestfold (Other); Helse Fonna (Other); Haukeland University Hospital (Other); Sykehuset Ostfold (Other); Helse Forde (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Åslaug Helland, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MATRIX-Rare
Record Dates: First submitted 2023-05-25; First posted 2023-11-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Rare Malignant Neoplasm
MeSH Terms: interventions — Imatinib Mesylate; trametinib; dabrafenib

STUDY DESIGN:
Intervention Model Description: simon two stage model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- treatment according to genetic alterations (Experimental): treatment according to genetic alterations
  Interventions: Drug: Imatinib; Drug: Trametinib; Drug: Dabrafenib

INTERVENTIONS:
Drug: Imatinib — imatinib treatment based on molecular alterations
Drug: Trametinib — According to biomarkers
Drug: Dabrafenib — According to biomarkers

SUMMARY:
Some rare cancers are hard-to-treat and patients have a poor prognosis. It is known that some of these patients have targetable molecular alterations, and some benefit from targeted drugs. However in many cases these drugs are not approved for the rare cancers.

In this study the aim is to do advanced molecular diagnostics to identify possible targets for therapy, and to treat accordingly.

DETAILED DESCRIPTION:
All patients will have the tumour cells diagnosed with a large genepanel, analyzing more than 500 genes on DNA / RNA level. Patients will be treated based on the molecular characteristics of the tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-2,
* identified biomarker,
* reasonable biochemistry

Exclusion Criteria:

* ECOG 3-5
* serious other diseases

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2033-11-30 (Estimated); Study Completion 2036-08-01 (Estimated)

PRIMARY OUTCOMES:
Radiological response evaluation at 16 weeks of treatment | 16 weeks
  Standard radiological response evaluation, like RECIST criteria.

SECONDARY OUTCOMES:
Molecular analyses predicting responses | 2 years
  Sequencing of tumor material and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Sigbjørn Smeland, MD PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No